CLINICAL TRIAL: NCT03822481
Title: Mindful Construal Diaries: Can the MCD Increase Mindfulness and Mindful Eating in Bariatric Surgery Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Birmingham City University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Bahia #004.17 BLSS FAEC; 226930 (Other: Human Research Authority (UK))
Record Dates: First submitted 2019-01-29; First posted 2019-01-30 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Obesity
Keywords: Post-Bariatric Surgery Weight-loss Diary
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: One group given the MCD (experimental) other group not given the MCD (control).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Participants in this arm were given the MCD. The MCD is a mindful eating intervention aimed at facilitating weight loss and cultivating a present centred awareness. The MCD consists of ten questions that an individual must consider while eating. Participants were required to consider the questions while eating (no writing required). Participants were asked to use the MCD at their three main meals (breakfast, lunch, dinner). The
  Interventions: Behavioral: Mindful Construal Diary
- Control (No Intervention): Participants in this arm were required to eat as normal and were not given the MCD until the study was complete.

INTERVENTIONS:
Behavioral: Mindful Construal Diary — A Mindful Eating Intervention
  Other Names: MCD
  Arms: Experimental

SUMMARY:
The study aims to test the Mindful Construal Diary (MCD- a mindful eating intervention) initially developed by Mantzios and Wilson. The diary aims to facilitate weight-loss, while also promoting a present centred awareness to current food consumption. There has yet to be any research testing the MCD in clinical populations.

DETAILED DESCRIPTION:
(BSP = Bariatric surgery patients) The MCD is an intervention that consists of 10 questions an individual must consider prior to eating, and revisit while eating. Mindfulness refers to being consciously aware in the present moment and being accepting to emotions, and in practice, ME can be defined as an awareness to thoughts, feelings and emotions related to current food consumption (e.g., portion size, feelings of hunger/satiety, and healthfulness of food). Being underpinned by both concepts, the MCD intervention prompts individuals to consider aspects of their meal by generating a more focused perspective to the experience of eating. Current applications of mindfulness in health-related settings are promising, benefits include long-term weight-loss, and decreases in symptoms associated with physical and psychiatric disorders. Although the MCD is similarly associated with weight-loss, existing literature on its utility within the bariatric surgery population is scant. Furthermore, as weight regain is often observed post-surgery, it is important to explore how the MCD can help BSP overcome this obstacles. Furthermore, as the MCD is yet to be applied to BSP, this research will also establish whether the MCD is effective in promoting mindfulness, ME and subsequent weight-loss in this population. The potential benefits of this research are broad, as it can help establish a novel approach to effective weight-loss in BSP, and equip health care practitioners with a cost-effective weight-loss intervention. This research will employ a mixed-method design, where participants will be asked to maintain use of the MCD when eating for a three month period, and at their usual care visit complete questionnaires and an interview. Participants will be recruited from Heartland Hospital's Bariatric Clinic.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or above
* Bariatric surgery patients cared for at Heartlands Hospital
* English speakers (reading and writing)
* Post bariatric surgery

Exclusion Criteria:

* Under the age of 18 years old
* A lack of capacity
* Not cared for at Heartlands Hospital
* Non-english speakers (reading and writing inc)
* Special communication needs
* Severe mental health illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
Weight loss | 3- months
  Weight loss - reduction in weight (kg) or body mass index (BMI)

SECONDARY OUTCOMES:
Mindfulness | 3- months
  Questionnaire - Five Facet Mindfulness Questionnaire - Short Form (FFMQ-SF; Bohlmeijer, Klooster, Fledderus, Veehof & Baer, 2011) is a 24-item measure which assesses five different but related aspects of mindfulness on a Likert scale, with a response scale of 1 (never or very rarely true) and 5 (very often or always true). Higher scores indicate higher levels of mindfulness (scores range from 24-120) total FFMQ scores are calculated by summing all items. The scale yields five subscales: observe, describe, acting with awareness, non-judgement and non-reactivity. Each subscales is calculated by summing each item that represents each subscale and subtracting six. Sample items include 'I tell myself that I shouldn't be feeling the way I'm feeling' and 'It seems I am running on automatic without much awareness of what I'm doing'. Higher scores are usually perceived positively as this represents engagement in positive practices which are associated with a range of health benefits.
Mindful eating | 3- months
  Questionnaire - Mindful Eating Scale (Hulbert-Williams, Joy & Hulbert-Williams 2013) is a 28-item measure which assesses mindful eating on a Likert scale, with a response scale of 1 (never) and 4 (usually). Higher scores indicate higher levels of mindful eating (scores range from 28-121), total Mindful Eating Scales scores are calculated by summing all items. The scale yields five subscales which assess different components of mindful eating: acceptance, awareness, non-reactivity, routine, distractibility and unstructured eating. Each subscales is calculated by summing each item that represents each subscale. Sample items include 'I criticise myself for the way I eat' and 'I notice how my food looks'. Higher scores are usually perceived positively as this represents engagement in positive eating practices.
Grazing | 3- months
  Questionnaire- The Grazing Scale (Lane & Szabo, 2013) is an 8-item measure which assesses an individual's tendency to eat small amounts of food, throughout the duration of the day, in a way which can be defined as unplanned, repetitious and uncontrolled. Responses are scored on a Likert scales 1 (rarely) and 4 (all of the time). Scores range from 8-32 and higher scores indicate higher levels of grazing, total scores are calculated by summing all items. Higher grazing scores are usually perceived as negative as this represents engagement in a maladaptive eating behaviour.
Eating Behaviours | 3- months
  Questionnaire - Dutch Eating Behaviour Questionnaire(DEBQ; Van Strien, 2002) is a 33-item scale which assesses eating behaviour styles. Responses are scored on a 5-point Likert scale (never-very often). Total scores range from 33-165, and higher scores relate to more engagement in maladaptive eating behaviours, total DEBQ scores are calculated by summing all items. The scale contains subscales which identify three different types of eating behaviours, these are: restrained, emotional, and external eating. Each subscales is calculated by summing each item that represents each subscale. Sample items include 'do you have the desire to eat when you are irritated?' and 'do you have the desire to eat when you are emotionally upset'.

CONTACTS AND LOCATIONS:
Locations (1):
- Heartlands Hospital, Birmingham, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data will not be shared outside of BCU.

REFERENCES:
- [Background] Mantzios M, Wilson JC. Making concrete construals mindful: a novel approach for developing mindfulness and self-compassion to assist weight loss. Psychol Health. 2014;29(4):422-41. doi: 10.1080/08870446.2013.863883. Epub 2013 Dec 4. PMID 24215123